CLINICAL TRIAL: NCT01883284
Title: Action of Epigenetic Modifiers in Cystic Fibrosis Treatment: ex Vivo Model of Nasal Epithelium of CF Patients
Brief Title: Action of Epigenetic Modifiers in Cystic Fibrosis Treatment
Acronym: Mod2EpiCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8870
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis; Healthy Subjects
Keywords: Cystic Fibrosis; nasal epithelia; mucins
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystic Fibrosis patients (CF) (Experimental): Tests in vitro after sampling nasal cells of CF patients or controls are the intervention done on these subjects
  Interventions: Other: Tests in vitro after sampling nasal cells of CF patients or controls
- Control subjects (non CF) (Other): Tests in vitro after sampling nasal cells of CF patients or controls are the intervention done on these subjects
  Interventions: Other: Tests in vitro after sampling nasal cells of CF patients or controls

INTERVENTIONS:
Other: Tests in vitro after sampling nasal cells of CF patients or controls — Nasal cells of CF patients or controls were collected by scratching of intermediate turbinate and cultured in vitro. Epigenetic modifiers treatment was applied to these ex vivo nasal epithelia. Then, mRNA, protein and secretions were quantified.

SUMMARY:
Epigenetic modifiers has been showed to rescue F508del-CFTR channel to apical membrane of epithelial cell lines. In this study, the investigators evaluate epigenetic modifiers effects firstly on CFTR rescue, then on secretion and synthesis of inflammatory factors (IL-8, LXA4 and SCGB1A1) and mucines (MUC5AC and MUC5B) in a dynamic epithelium model using an air-liquide interface culture of nasals cells from CF patients or controls.

ELIGIBILITY:
General inclusion criteria :

* informed consent
* benefit from disease insurance regimen
* men and women

Inclusion Criteria for CF patients

* 2 severe CF mutations
* age superior or equal to 12

Inclusion Criteria for controls :

* age superior or equal to 18
* no smoker (for 5 years)

General exclusion criteria :

* participation to an other interventionnal study
* subject in exclusion period
* law protected subject
* pregnant and breast fooding

Specific Exclusion Criteria:

* Xylocaine hypersensibility
* Porphyria
* severe hepatic failure
* Epilepsy
* Severe cardiac failure
* local anesthesic contra indication

Specific Control subject Exclusion Criteria:

* respiratory disease
* cystic fibrosis
* acute infection < 6 weeks
* on treatment
* antibiotic treatment < 3 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mature CFTR protein percentage variation after in vitro epigenetics modifiers treatment | 24 months

SECONDARY OUTCOMES:
Pro-inflammatory cytokines number variations after epigenetic modifiers treatment | 24 months
Anti-inflammatory cytokines number variations after epigenetic modifiers treatment | 24 months
Mucin composition variations after epigenetic modifiers treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël RC CHIRON, MD, Principal Investigator — Arnaud de Villeneuve CHU Montpellier
Locations (1):
- Respiratory Diseases Department, Montpellier, France